CLINICAL TRIAL: NCT03288974
Title: Post Marketing Surveillance on Safety Evaluation of POMALYST® (Pomalidomide) Treatment of Multiple Myeloma in Korea
Acronym: Pomalyst PMS
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NIPMS-POM-KR-001; U1111-1201-1712 (Registry Identifier: WHO)
Record Dates: First submitted 2017-09-05; First posted 2017-09-20 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; POMALYST®; Pomalidomide; Observational; Korea; Post Marketing Surveillance[PMS]; Relapsed and Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — pomalidomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Post Marketing Survey of MM patients treated with POMALYST®: As a method of POMALYST® PMS, Drug Use Examination (DUE) is planned and designed to comply with the regulatory requirement in consequence of approval of a new drug in Korea. This DUE is a non-interventional, observational and post-marketing surveillance, which is conducted as a regulatory required procedure to evaluate product safety of a new drug treatment in clinical routine practice in Korea. And this DUE will be conducted in compliance with the local guideline [standard for Re-examination of New Drugs, etc.] as a post approval commitment.
  Interventions: Drug: POMALYST® (Pomalidomide)

INTERVENTIONS:
Drug: POMALYST® (Pomalidomide) — The recommended starting dose of POMALYST is 4 mg once daily taken orally on Days 1 to 21 of repeated 28-day cycles. The recommended dose of dexamethasone is 40 mg orally once daily on Days 1, 8, 15 and 22 of each 28-day treatment cycle

SUMMARY:
PMS period: 09Jun2017 ~ 08Jun2023 Target no.: 600patients

indication: POMALYST in combination with dexamethasone is indicated in the treatment of patients with relapsed and refractory multiple myeloma who have received at least two prior treatment regimens, including both lenalidomide and bortezomib

The primary objective of this Drug Use Examination (DUE) is to evaluate safety of POMALYST® (Pomalidomide) treatment of multiple myeloma in the clinical routine practice in Korea.

The secondary objective of this DUE is to evaluate effectiveness of POMALYST® (Pomalidomide) treatment of multiple myeloma in the clinical routine practice in Korea.

ELIGIBILITY:
Inclusion Criteria:

The main criteria for inclusion of this DUE is the same as the approved package insert of POMALYST® in Korea. Based on the current PI, patients who are treated with POMALYST® based on the following criteria, can be registered into this DUE.

* POMALYST® in combination with dexamethasone is indicated in the treatment of patients with relapsed and refractory multiple myeloma who have received at least two prior treatment regimens, including both lenalidomide and bortezomib.

The actual inclusion criteria and patient population who can start with POMALYST® treatment will be narrowed down according to the local health insurance reimbursement condition.

Exclusion Criteria:

* There's no exclusion criteria

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are treated with POMALYST® based on the following criteria, can be registered into this DUE.
  •POMALYST® in combination with dexamethasone is indicated in the treatment of patients with relapsed and refractory multiple myeloma who have received at least two prior treatment regimens, including both lenalidomide and bortezomib.
Sampling Method: Non-Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
Adverse events | From enrollment until at least 28 days after completion of study treatment
  Any untoward medical occurrence in a patient administered a medicinal product and which does not necessarily have a causal relationship with this treatment, i.e., any unfavorable and unintended sign (e.g. an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product whether or not considered related to the medicinal product.se temporally associated with the use of a medicinal product whether or not considered related to the medicinal product.

SECONDARY OUTCOMES:
Overall response rate | Up to approximately 5.6 months
  The percentage of patients who achieve CR (complete response), sCR (stringent complete response), Immunophenotypic CR, Molecular CR, VGPR (very good partial response) and PR (partial response) will be evaluated as overall response rate during POMALYST® treatment period based on International Myeloma Working Group Criteria for Multiple Myeloma.
  Analysis and reporting for efficacy will be done at every 6months for the first 2years and after then, annual report(3,4,5th yearly report) and CSR for all data of 6years will be submitted to MFDS in accordance with MFDS guideline.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (33):
- South Korea (33):
  - Korea University Ansan Hospital, Ansan
  - Hallym University Sacred Heart Hospital, Anyang
  - Soonchunhyang University Hospital, Bucheon-si
  - Inje University Busan Paik Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Keimyung University Dongsan Medical, Daegu
  - Yeungnam University Medical Center, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Local Institution - 021, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hwasun Hospital, Hwasun
  - Inha University Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Local Institution - 024, Jinju
  - Inje University Sanggye Paik Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The catholic University of Korea Seoul St. Maty's, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - Ewha Womans University Medical, Seoul
  - Korea University Guro Hospital, Seoul
  - Local Institution - 001, Seoul
  - Local Institution - 002, Seoul
  - Ajou Unversity Medical Center, Suwon
  - Ulsan University Hospital, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju
  - Pusan National University Yangsan, Yangsan